CLINICAL TRIAL: NCT07204561
Title: Analysis of the CeraVe Emollient Effect on Restoring the Hydration of the Skin Barrier as Maintenance Regimen in Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: CeraVe Effect on Restoring Skin Hydration as Maintenance Regimen in Subjects With Mild to Moderate Atopic Dermatitis
Acronym: DA_CeraVe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SID05
Record Dates: First submitted 2025-06-09; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: A clinical assessment of disease severity (EASI) will be conducted at three separate visits: a screening visit on Day -15, and two visits on Days 1 and 42. At the screening visit, subjects will be given a medical corticosteroid topical treatment (mometasone furoate cream) to improve their EASI score by at least 90% between Day -15 and Day 1. Only individuals with an EASI score reduction of at least 90% between Day -15 and Day 1 will be randomised into two groups. Group 1 will enter the maintenance phase with CeraVe emollient, while group 2 will be treated with a standard emollient. Both groups will be provided with a basic detergent for washing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - CeraVe (Experimental): Subjects who agree to participate in this study and have previously signed a specific informed consent form will enter the maintenance phase with CeraVe emollient following corticosteroid treatment as per clinical practice.
  Interventions: Other: CeraVe Moisturizing Cream
- Arm 2 - Galenico (Active Comparator): Subjects who agree to participate in this study and have previously signed a specific informed consent form will enter the maintenance phase with a common soft emollient after corticosteroid treatment, as per clinical practice.
  Interventions: Other: Galenico

INTERVENTIONS:
Other: CeraVe Moisturizing Cream — During the 42-day maintenance phase, subjects must apply the CeraVe emollient twice a day after washing with the basic detergent as part of their normal hygiene routine.
  Arms: Arm 1 - CeraVe
Other: Galenico — During the 42-day maintenance phase, subjects must apply the emollient twice a day after washing with the basic detergent as part of their normal hygiene routine.
  Arms: Arm 2 - Galenico

SUMMARY:
This is an open-label, randomised, comparative, prospective, interventional study of a cosmetic product.

DETAILED DESCRIPTION:
Atopic dermatitis is a common chronic inflammatory skin condition that affects individuals with specific alterations to the epidermal barrier. It is also characterised by defective ceramide production. Emollients play an important role in managing atopic dermatitis, including during the maintenance phase following topical cortisone therapy. However, the effect of CeraVe emollient cream on restoring skin barrier hydration has yet to be investigated.

The primary objective is to evaluate the effect of the CeraVe emollient on restoring skin barrier hydration as a maintenance regimen in subjects with mild to moderate atopic dermatitis. The secondary objectives are to evaluate and compare the cosmetic acceptability of CeraVe with that of a commonly used emollient produced in a licensed pharmacy laboratory, and to assess the differences in ADCT (Atopic Dermatitis Control Tool) scores between groups.

Subjects with mild-to-moderate atopic dermatitis (AD), as defined by an EASI score of 1-21, will be enrolled in the study. Only individuals with an EASI score reduction of at least 90% between screening (Day -15) and Visit 1 (Day 1) will be randomised into two groups. Group 1 will enter the maintenance phase with CeraVe emollient, while group 2 will be treated with a standard emollient. Both groups will be provided with a basic detergent for washing.

If the participant experiences a relapse of atopic dermatitis (AD), as reported in their diary and in the eCRF, they should discontinue the application of CeraVe Emollient or a common soft emollient. The subject should be examined by a physician and treated according to the severity of the AD. In this case, they will be withdrawn from the study.

ELIGIBILITY:
Inclusion criteria:

Subjects with clinically confirmed mild-to-moderate atopic dermatitis (AD), as defined by an Eczema Area and Severity Index (EASI) score of 1-21, whose lesions will clear after treatment with a steroid and who will experience at least a 90% reduction in their EASI score.

- Participants of any gender, aged 18 years or over, from any phototype or ethnic group.

Participants must be willing and able to give informed consent to participate in the study.

Exclusion criteria:

* Age <18 years. Participants who are unwilling or unable to give informed consent to participate in the study.
* Receiving any systemic treatment for atopic dermatitis (AD), including corticosteroids, cyclosporine, any approved biologics or JAK inhibitors.
* Any dermatological disorder which, in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics (except AD).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in EASI score | From enrollment to the end of treatment at 6 weeks
  Changes in EASI (Eczema Area and Severity Index) score. A clinical assessment of disease severity (EASI) will be conducted at three separate visits: a screening visit on Day -15, and two visits on Days 1 and 42. At the screening visit, subjects will be given a medical corticosteroid topical treatment (mometasone furoate cream) to improve their EASI score by at least 90% between Day -15 and Day 1. Only individuals with an EASI score reduction of at least 90% between Day -15 and Day 1 will be randomised into two groups. EASI score interpretation: 0: clear; 0.1-1: almost clear; 1.1-7: mild; 7.1-21: moderate; 21.1-50: severe; 50.1-72: very severe.

SECONDARY OUTCOMES:
Cosmetic acceptability | From visit 1 to the end of treatment at 6 weeks
  The cosmetic acceptability of the emollients is assessed in two groups of participants using specific questionnaires. The 21 questions covered texture, fluidity and penetration of the emollients. Scoring was as follows: 0 = totally agree; 1 = agree; 2 = disagree; 3 = totally disagree.
Changes in ADCT score | From enrollment to the end of treatment at 6 weeks
  The ADCT (Atopic Dermatitis Control Tool) score is compared between groups. This is a set of six concise questions designed to evaluate the various aspects of atopic dermatitis (AD) control that have been identified as important by patients and clinicians. Each question is scored between 0 and 4 points (0 = none, 4 = very severe). The sum of the points from the answers to the six ADCT questions is the ADCT total score. The ADCT total score will be between 0 and 24.
The number and proportion of subjects who experience a relapse of AD. | From enrollment to the end of treatment at 6 weeks
  The number and proportion of subjects who experience a relapse of atopic dermatitis (AD) in the two groups. If a relapse of AD occurs, the subject should discontinue the application of the CeraVe emollient or the common soft emollient. They should be examined by a physician and treated according to the severity of the AD. In this case, they will be withdrawn from the study.
Changes in the visual appearance of the skin barrier over time, as observed by comparing images collected during the three scheduled study visits. | From enrollment to the end of treatment at 6 weeks
  We will compare images of visual changes to the skin barrier collected at screening and visits 1 and 42. The images will only refer to areas affected by the disease and will not contain any recognisable features that could identify the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione PTV - Policlinico Tor Vergata, Roma, RM, Italy